CLINICAL TRIAL: NCT06565715
Title: Effect of Remazolam on Hemodynamics During Hepatectomy Under General Anesthesia Combined With Thoracic Epidural Anesthesia
Brief Title: Effect of Remazolam on Hemodynamics During Hepatectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jun Zhang (Other)
Responsible Party: Sponsor-Investigator, Jun Zhang, Professor, Fudan University
Organization: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Remazolam-Hepatectomy
Record Dates: First submitted 2024-08-16; First posted 2024-08-22 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2024-08

CONDITIONS: Hemodynamic Instability
MeSH Terms: interventions — remimazolam; Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remazolam group (Experimental): Remazolam group: remazolam is administered 0.3mg/kg intravenous for anesthesia induction.
  Interventions: Drug: Remimazolam
- Propofol group (Other): Propofol group: propofol is administered 2mg/kg intravenous for anesthesia induction.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Remimazolam — Remimazolam is used for sedation during anesthetic induction and maintenance.
  Other Names: rebenin
  Arms: Remazolam group
Drug: Propofol — propofol is used for sedation during anesthetic induction and maintenance.
  Other Names: Propofol emulsion
  Arms: Propofol group

SUMMARY:
There is high incidence of hemodynamic instability in patients undergoing hepatectomy with low central venous pressure, especially in general anesthesia combined with epidural anesthesia. Remazolam, a new benzodiazepine, has no significant cardiovascular inhibitory effect. Investigators hypothesis that remazolam will provide better hemodynamic when compared with propofol in patients undergoing hepatectomy with general anesthesia combined with epidural anesthesia.

DETAILED DESCRIPTION:
Investigators plan to adopt the following strategies in the clinical study of this project: (1) To compare remazolam and propofol during anesthetic induction and maintenance; (2) Remazolam group: remazolam is administered 0.3mg/kg intravenous for anesthesia induction. Propofol group: propofol is administered 2mg/kg intravenous for anesthesia induction; (3) Epidural analgesia is used during perioperative period, and remifentanil pump injection is used during the operation to assist the subjects to tolerate the tracheal catheter; (4) the haemodynamic instability score (Hemodynamic instability score) is used to comprehensively evaluate intraoperative hemodynamic status. (5) To evaluate the incidence of postoperative complications. Through the above strategies, investigators further determine the optimization effect of remazolam, a novel benzodiazepine drug, on intraoperative hemodynamics in patients undergoing low central venous pressure hepatectomy, and further lay an empirical foundation for the routine use of remazolam in clinical hepatectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who sign informed consent and are willing to complete the study according to the plan;
2. Over 18 years of age;
3. ASA grade Ⅰ ~ Ⅲ;
4. Elective surgery;
5. General anesthesia combined with epidural anesthesia;
6. Child Pugh is classified as Level A

Exclusion Criteria:

1. Abnormal coagulation function;
2. Abnormal platelet;
3. A history of drug dependence;
4. Neurological diseases;
5. Severe sinus bradycardia (HR<50 beats/min);
6. Atrial fibrillation;
7. Systolic blood pressure ≥200mmHg and/or diastolic blood pressure ≥120mmHg.
8. Cardiac insufficiency.
9. Child Pugh is classified as B or C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-08-23 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-11-08 (Actual)

PRIMARY OUTCOMES:
Hemodynamic instability score | intraoperative
  The hemodynamic instability score is calculated as a weighted continuous measure ranging from 0 to 160 points, intended to reflect deviations of blood pressure and heart rate from predefined thresholds, and infusion rates of vasoactive agents and fluids.

SECONDARY OUTCOMES:
Cardiac index （CI） | intraoperative
  The parameter of CI is measured by advanced hemodynamic monitoring device.
Stroke volume variation (SVV) | intraoperative
  The parameter of SVV is measured by advanced hemodynamic monitoring device.
Systemic vascular resistance index (SVRI) | intraoperative
  The parameter of SVRI is measured by advanced hemodynamic monitoring device.
Complications in 1 week after surgery | 1 week after surgery
  Complications occured within 1 week after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, Professor, Study Chair — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
The data sets are available from the corresponding author on reasonable request.

REFERENCES:
- [Derived] Qian Y, Hou W, Yang L, Chen N, Zhang J. A randomized trial evaluating hemodynamics during minor hepatectomy under general anesthesia combined with thoracic epidural anesthesia: remimazolam versus propofol. BMC Anesthesiol. 2025 Aug 20;25(1):413. doi: 10.1186/s12871-025-03290-w. PMID 40836208